CLINICAL TRIAL: NCT02345629
Title: Minimally Invasive Cordotomy for Refractory Cancer Pain
Brief Title: Cordotomy for Refractory Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0833; NCI-2015-00206 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Advanced Cancers; Pain
Keywords: Refractory cancer pain; Cordotomy; Sharpness pain sensory testing; Heat pain sensory testing; Symptom questionnaire; Advanced cancers; Pain
MeSH Terms: conditions — Pain; Cancer Pain | interventions — Cordotomy; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cordotomy Group (Experimental): Radiologist performs a spinal tap to inject a contrast drug into the spinal fluid. A 20G spinal needle guided by real-time CT scan to the C1-C2 level opposite to participant's pain. A radiofrequency electrode inserted through the spinal needle into the spinal cord, to the anatomic location of the spinothalamic tract. Once ideal position of the electrode is confirmed, 1 or 2 radiofrequency ablations performed at 70C-80C for 60 seconds. The procedure will take 1-2 hours. Quantitative sensory testing on day prior to procedure, and on postoperative days number 1 and 7. Pain and symptom questionnaire completed at baseline, over the phone during the first week of study, and at each follow up visit/phone call. Participants undergo quantitative sensory testing on day prior to procedure, and on postoperative days number 1 and 7. Sensory testing to include sharpness and heat detection.
  Interventions: Procedure: Cordotomy; Behavioral: Pain/Symptom Questionnaire; Procedure: Sharpness Sensory Testing; Procedure: Heat Pain Sensory Testing
- Comprehensive Medical Management Group (Active Comparator): Participants receive best supportive care for 1 week. Depending on pain level after the first week, they may have a cordotomy at that time. Pain and symptom questionnaire completed at baseline, over the phone during the first week of study, and at each follow up visit/phone call.
  Interventions: Procedure: Cordotomy; Procedure: Sharpness Sensory Testing; Procedure: Heat Pain Sensory Testing

INTERVENTIONS:
Procedure: Cordotomy — Radiologist performs a spinal tap to inject a contrast drug into the spinal fluid. A 20G spinal needle guided by real-time CT scan to the C1-C2 level opposite to participant's pain. A radiofrequency electrode inserted through the spinal needle into the spinal cord, to the anatomic location of the spinothalamic tract. Once ideal position of the electrode is confirmed, 1 or 2 radiofrequency ablations performed at 70C-80C for 60 seconds. The procedure will take 1-2 hours.
Behavioral: Pain/Symptom Questionnaire — Pain and symptom questionnaire completed at baseline, by phone during first week of study, and once each month by phone during 6 month follow up.
  Other Names: Survey
  Arms: Cordotomy Group
Procedure: Sharpness Sensory Testing — Sharpness detection determined using 8, 10, 16, 20, 32, 64, and 128g weighted needle devices. Each stimulus applied for about 1 second in ascending order. Participants asked to rate each stimulus as producing the sensation of touch, pressure, sharp, or pain. The sharpness detection threshold defined as the mean force of the stimuli deemed ''sharp'' or ''painful'' from 3 trials separated by an average interval of 30 to 90 seconds.
Procedure: Heat Pain Sensory Testing — Thermal ramps will applied using a 3.6 x 3.6 cm Peltier thermode (Medoc Inc.) from a baseline temperature set at 32C. Skin heated at a rate of 0.30C/s, and participants asked to signal when the stimulus is perceived as first becoming warmer and then painfully hot.

SUMMARY:
The goal of this clinical research study is to learn if a cordotomy reduces pain in patients with unmanageable cancer pain. A cordotomy is a procedure, guided by computed tomography (CT) scans, that is performed on the spinal cord and is designed to reduce pain transmission.

DETAILED DESCRIPTION:
Baseline Tests:

If you agree to take part in this study, you will have the following tests and procedures:

* You will have a physical exam.
* You will complete 2 questionnaires that ask about any symptoms and pain you may be having. It should take about 10 minutes to complete the questionnaires.
* You will have sensory testing. These are tests to measure your level of pain and feelings of hot and cold in the foot, palm of the hand, and the area where your pain is the worst.

Study Groups:

You will be assigned to 1 of 2 groups. You will have an equal chance of being in either group.

* If you are in Group 1, you will have a cordotomy the day after the baseline tests.
* If you are in Group 2, you will receive the best supportive care for 1 week. Depending on your pain level after the first week, you may have a cordotomy at that time.

Cordotomy Procedure:

If you are in Group 2, you will have a physical exam on the day of the cordotomy.

The cordotomy procedure will take place in the CT scan area. Before the procedure, a radiologist will perform a spinal tap to inject a contrast drug into the spinal fluid. This will allow researchers to see the spinal cord well on the CT scan. You will be taken to the diagnostic CT scanner and given local anesthetic and standard drugs by vein to help you feel comfortable. A needle will be inserted using CT scan guidance into the side of the neck opposite to your pain. A radiofrequency electrode will pass through the needle into your spinal cord, and your nerve reactions to movement and sensation will be checked. If these reactions are not satisfactory, the needle will be adjusted or the procedure will be stopped.

Once the best position for the needle is found, the surgeon will use the radiofrequency electrode to heat the pain pathway in the spinal cord at that point, so that your sensation of pain is less. During this process, you will be checked for signs of weakness.

The procedure will take 1-2 hours. You will sign a separate consent form for this procedure.

One day to one week after the procedure, you will have a MRI to help determine the effect of the cordotomy on your spinal nerves.

Study Tests and Phone Calls:

All participants will return to the clinic or be seen in the hospital the day after the cordotomy and again 1 week later. At these visits, you will have a physical exam and sensory testing.

You will be called by phone 1 time during the first week of the study. You will be asked to complete the pain and symptom questionnaires over the phone. If you are not able to return to the clinic a week after your cordotomy, you will also be called at that time.

Follow-Up Calls:

You will return to the clinic or be called on the phone 1 time each month for as long as you are still having pain. You will be asked to complete the pain and symptom questionnaires.

Length of Study Participation:

You active participation in this study will be over 6 months after your cordotomy, if you have one.

This is an investigational study. It is investigational to perform a cordotomy to learn if the procedure reduces pain in patients with unmanageable cancer pain.

Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with one-sided, somatic pain due to tumor involvement below the shoulder level (C5 dermatome).
2. Patients with refractory cancer pain who are seen by the Supportive Care or Pain Medicine teams, and who either (1) are on appropriate opioid therapy at the time of consultation, or (2) who undergo an initial consultation and at least 2 clinical follow-up evaluations by these services.
3. Patients with a life expectancy greater than 1 month.
4. Patients must be 18 years old or older.
5. Patients must be able to read, speak and understand English or Spanish.

Exclusion Criteria:

1) Patients with significant pulmonary dysfunction, large intracranial metastases, or significant thrombocytopenia (platelet count refractory to transfusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-03-10 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity using a 0-10 numeric rating scale | Day 1 and Day 8
  The response rate for both the cordotomy and control groups determined by the change in pain intensity between day 1 and day 8. Pain intensity assessed before and after cordotomy using a 0-10 numeric rating scale. Response rate defined as a 33% reduction in pain intensity with a 95% confidence interval, separately within each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Viswanathan, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org